CLINICAL TRIAL: NCT04891055
Title: Prospective Translational Study Investigating Predictors of Outcome in Metastatic Renal Cell Carcinoma Patients Treated With Nivolumab (I-Rene Trial)
Acronym: I-Rene
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Fondazione IRCCS Istituto Nazionale dei Tumori, Milano (Other)
Collaborators: Ministero della Salute, Italy (Other)
Responsible Party: Sponsor
Other Study IDs: INT 71/18
Record Dates: First submitted 2021-05-07; First posted 2021-05-18 (Actual); Last update posted 2021-05-18 (Actual); Status verified 2021-05

CONDITIONS: Metastatic Renal Cell Carcinoma
Keywords: Metastatic renal cell carcinoma; Predictive factors
MeSH Terms: conditions — Carcinoma, Renal Cell

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- patients treated with nivolumab: Patients candidates for II line therapy with Nivolumab from clinical practice
- patients treated with TKI: Patients candidates for II line therapy with TKI from clinical practice

SUMMARY:
Prospective translational study investigating predictors of outcome in metastatic renal cell carcinoma patients treated with Nivolumab (I-Rene trial)

DETAILED DESCRIPTION:
Prospective translational study investigating predictors of outcome in metastatic renal cell carcinoma patients treated with Nivolumab (I-Rene trial)

ELIGIBILITY:
Inclusion Criteria:

* Written informed consent
* metastatic renal cell carcinoma (a clear-cell/ not clear-cell)
* Progression to previous treatment with tyrosine kinase inhibitors
* Patients candidates for II-line therapy with Nivolumab (or tyrosine kinase inhibitors-in the control arm)

Exclusion Criteria:

none

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: metastatic renal cell carcinoma
Sampling Method: Non-Probability Sample
Enrollment: 90 (Estimated)
Dates: Start 2018-11-29 (Actual); Primary Completion 2021-11-29 (Estimated); Study Completion 2021-11-29 (Estimated)

PRIMARY OUTCOMES:
Investigate the predictive role of circulating miRNAs will be studied with OpenArray technology (OA, Thermo Fisher) | 36 months
  To investigate the predictive role of circulating miRNAs in patients who respond to nivolumab versus those who do not respond before treatment, after two infusions (4 weeks), at the first radiological re-evaluation (12 weeks) and at the time of disease progression.
To evaluate whether the immunological profile of tumor tissue or circulating tumor cells Using Multiplexed Biomarker Imaging (MBI), multiparametric flow cytometry | 36 months
  To evaluate whether the immunological profile of tumor tissue or circulating tumor cells may be a potential predictor of clinical response in patients treated with nivolumab. Using Multiplexed Biomarker Imaging (MBI), multiparametric flow cytometry
Characterize alterations in genes and signal transmission pathways. Using Next Generation Sequencing, NGS) | 36 months
  o characterize alterations in genes and signaling pathways and to identify mutational burden differences between tumors of patients with metastatic renal cell carcinoma who respond or not to nivolumab.

CONTACTS AND LOCATIONS:
Overall Officials: Giuseppe Procopio, MD, Principal Investigator — Fondazione IRCCS Istituto Nazionale Tumori Milano
Locations (1):
- Fondazione IRCCS Istituto Nazionale Tumori, Milan, Italy

REFERENCES:
- [Background] Motzer RJ, Escudier B, McDermott DF, George S, Hammers HJ, Srinivas S, Tykodi SS, Sosman JA, Procopio G, Plimack ER, Castellano D, Choueiri TK, Gurney H, Donskov F, Bono P, Wagstaff J, Gauler TC, Ueda T, Tomita Y, Schutz FA, Kollmannsberger C, Larkin J, Ravaud A, Simon JS, Xu LA, Waxman IM, Sharma P; CheckMate 025 Investigators. Nivolumab versus Everolimus in Advanced Renal-Cell Carcinoma. N Engl J Med. 2015 Nov 5;373(19):1803-13. doi: 10.1056/NEJMoa1510665. Epub 2015 Sep 25. PMID 26406148
- [Background] Rizvi NA, Hellmann MD, Snyder A, Kvistborg P, Makarov V, Havel JJ, Lee W, Yuan J, Wong P, Ho TS, Miller ML, Rekhtman N, Moreira AL, Ibrahim F, Bruggeman C, Gasmi B, Zappasodi R, Maeda Y, Sander C, Garon EB, Merghoub T, Wolchok JD, Schumacher TN, Chan TA. Cancer immunology. Mutational landscape determines sensitivity to PD-1 blockade in non-small cell lung cancer. Science. 2015 Apr 3;348(6230):124-8. doi: 10.1126/science.aaa1348. Epub 2015 Mar 12. PMID 25765070
- [Background] Cancer Genome Atlas Research Network. Comprehensive molecular characterization of clear cell renal cell carcinoma. Nature. 2013 Jul 4;499(7456):43-9. doi: 10.1038/nature12222. Epub 2013 Jun 23. PMID 23792563
- [Background] Hakimi AA, Ostrovnaya I, Reva B, Schultz N, Chen YB, Gonen M, Liu H, Takeda S, Voss MH, Tickoo SK, Reuter VE, Russo P, Cheng EH, Sander C, Motzer RJ, Hsieh JJ; ccRCC Cancer Genome Atlas (KIRC TCGA) Research Network investigators. Adverse outcomes in clear cell renal cell carcinoma with mutations of 3p21 epigenetic regulators BAP1 and SETD2: a report by MSKCC and the KIRC TCGA research network. Clin Cancer Res. 2013 Jun 15;19(12):3259-67. doi: 10.1158/1078-0432.CCR-12-3886. Epub 2013 Apr 25. PMID 23620406
- [Background] Pena-Llopis S, Vega-Rubin-de-Celis S, Liao A, Leng N, Pavia-Jimenez A, Wang S, Yamasaki T, Zhrebker L, Sivanand S, Spence P, Kinch L, Hambuch T, Jain S, Lotan Y, Margulis V, Sagalowsky AI, Summerour PB, Kabbani W, Wong SW, Grishin N, Laurent M, Xie XJ, Haudenschild CD, Ross MT, Bentley DR, Kapur P, Brugarolas J. BAP1 loss defines a new class of renal cell carcinoma. Nat Genet. 2012 Jun 10;44(7):751-9. doi: 10.1038/ng.2323. PMID 22683710
- [Background] Brooks SA, Brannon AR, Parker JS, Fisher JC, Sen O, Kattan MW, Hakimi AA, Hsieh JJ, Choueiri TK, Tamboli P, Maranchie JK, Hinds P, Miller CR, Nielsen ME, Rathmell WK. ClearCode34: A prognostic risk predictor for localized clear cell renal cell carcinoma. Eur Urol. 2014 Jul;66(1):77-84. doi: 10.1016/j.eururo.2014.02.035. Epub 2014 Feb 25. PMID 24613583
- [Background] Tumeh PC, Harview CL, Yearley JH, Shintaku IP, Taylor EJ, Robert L, Chmielowski B, Spasic M, Henry G, Ciobanu V, West AN, Carmona M, Kivork C, Seja E, Cherry G, Gutierrez AJ, Grogan TR, Mateus C, Tomasic G, Glaspy JA, Emerson RO, Robins H, Pierce RH, Elashoff DA, Robert C, Ribas A. PD-1 blockade induces responses by inhibiting adaptive immune resistance. Nature. 2014 Nov 27;515(7528):568-71. doi: 10.1038/nature13954. PMID 25428505
- [Background] Rosenberg JE, Hoffman-Censits J, Powles T, van der Heijden MS, Balar AV, Necchi A, Dawson N, O'Donnell PH, Balmanoukian A, Loriot Y, Srinivas S, Retz MM, Grivas P, Joseph RW, Galsky MD, Fleming MT, Petrylak DP, Perez-Gracia JL, Burris HA, Castellano D, Canil C, Bellmunt J, Bajorin D, Nickles D, Bourgon R, Frampton GM, Cui N, Mariathasan S, Abidoye O, Fine GD, Dreicer R. Atezolizumab in patients with locally advanced and metastatic urothelial carcinoma who have progressed following treatment with platinum-based chemotherapy: a single-arm, multicentre, phase 2 trial. Lancet. 2016 May 7;387(10031):1909-20. doi: 10.1016/S0140-6736(16)00561-4. Epub 2016 Mar 4. PMID 26952546
- [Background] Gerlinger M, Horswell S, Larkin J, Rowan AJ, Salm MP, Varela I, Fisher R, McGranahan N, Matthews N, Santos CR, Martinez P, Phillimore B, Begum S, Rabinowitz A, Spencer-Dene B, Gulati S, Bates PA, Stamp G, Pickering L, Gore M, Nicol DL, Hazell S, Futreal PA, Stewart A, Swanton C. Genomic architecture and evolution of clear cell renal cell carcinomas defined by multiregion sequencing. Nat Genet. 2014 Mar;46(3):225-233. doi: 10.1038/ng.2891. Epub 2014 Feb 2. PMID 24487277
- [Background] Filipazzi P, Valenti R, Huber V, Pilla L, Canese P, Iero M, Castelli C, Mariani L, Parmiani G, Rivoltini L. Identification of a new subset of myeloid suppressor cells in peripheral blood of melanoma patients with modulation by a granulocyte-macrophage colony-stimulation factor-based antitumor vaccine. J Clin Oncol. 2007 Jun 20;25(18):2546-53. doi: 10.1200/JCO.2006.08.5829. PMID 17577033
- [Background] Walter S, Weinschenk T, Stenzl A, Zdrojowy R, Pluzanska A, Szczylik C, Staehler M, Brugger W, Dietrich PY, Mendrzyk R, Hilf N, Schoor O, Fritsche J, Mahr A, Maurer D, Vass V, Trautwein C, Lewandrowski P, Flohr C, Pohla H, Stanczak JJ, Bronte V, Mandruzzato S, Biedermann T, Pawelec G, Derhovanessian E, Yamagishi H, Miki T, Hongo F, Takaha N, Hirakawa K, Tanaka H, Stevanovic S, Frisch J, Mayer-Mokler A, Kirner A, Rammensee HG, Reinhardt C, Singh-Jasuja H. Multipeptide immune response to cancer vaccine IMA901 after single-dose cyclophosphamide associates with longer patient survival. Nat Med. 2012 Aug;18(8):1254-61. doi: 10.1038/nm.2883. Epub 2012 Jul 29. PMID 22842478
- [Background] Verderio P, Bottelli S, Ciniselli CM, Pierotti MA, Gariboldi M, Pizzamiglio S. NqA: an R-based algorithm for the normalization and analysis of microRNA quantitative real-time polymerase chain reaction data. Anal Biochem. 2014 Sep 15;461:7-9. doi: 10.1016/j.ab.2014.05.020. Epub 2014 Jun 2. PMID 24892985
- [Background] Verderio P, Bottelli S, Pizzamiglio S, Ciniselli CM. Developing miRNA signatures: a multivariate prospective. Br J Cancer. 2016 Jun 28;115(1):1-4. doi: 10.1038/bjc.2016.164. No abstract available. PMID 27351381
- [Background] Hugo W, Zaretsky JM, Sun L, Song C, Moreno BH, Hu-Lieskovan S, Berent-Maoz B, Pang J, Chmielowski B, Cherry G, Seja E, Lomeli S, Kong X, Kelley MC, Sosman JA, Johnson DB, Ribas A, Lo RS. Genomic and Transcriptomic Features of Response to Anti-PD-1 Therapy in Metastatic Melanoma. Cell. 2016 Mar 24;165(1):35-44. doi: 10.1016/j.cell.2016.02.065. Epub 2016 Mar 17. PMID 26997480
- [Background] Zhou L, Liu XD, Sun M, Zhang X, German P, Bai S, Ding Z, Tannir N, Wood CG, Matin SF, Karam JA, Tamboli P, Sircar K, Rao P, Rankin EB, Laird DA, Hoang AG, Walker CL, Giaccia AJ, Jonasch E. Targeting MET and AXL overcomes resistance to sunitinib therapy in renal cell carcinoma. Oncogene. 2016 May;35(21):2687-97. doi: 10.1038/onc.2015.343. Epub 2015 Sep 14. PMID 26364599
- [Background] Gabrilovich DI, Ostrand-Rosenberg S, Bronte V. Coordinated regulation of myeloid cells by tumours. Nat Rev Immunol. 2012 Mar 22;12(4):253-68. doi: 10.1038/nri3175. PMID 22437938
- [Background] Geissler K, Fornara P, Lautenschlager C, Holzhausen HJ, Seliger B, Riemann D. Immune signature of tumor infiltrating immune cells in renal cancer. Oncoimmunology. 2015 Feb 3;4(1):e985082. doi: 10.4161/2162402X.2014.985082. eCollection 2015 Jan. PMID 25949868
- [Background] Gebhardt C, Sevko A, Jiang H, Lichtenberger R, Reith M, Tarnanidis K, Holland-Letz T, Umansky L, Beckhove P, Sucker A, Schadendorf D, Utikal J, Umansky V. Myeloid Cells and Related Chronic Inflammatory Factors as Novel Predictive Markers in Melanoma Treatment with Ipilimumab. Clin Cancer Res. 2015 Dec 15;21(24):5453-9. doi: 10.1158/1078-0432.CCR-15-0676. Epub 2015 Aug 19. PMID 26289067
- [Background] Hammers HJ, Plimack ER, Infante JR, Rini BI, McDermott DF, Lewis LD, Voss MH, Sharma P, Pal SK, Razak ARA, Kollmannsberger C, Heng DYC, Spratlin J, McHenry MB, Amin A. Safety and Efficacy of Nivolumab in Combination With Ipilimumab in Metastatic Renal Cell Carcinoma: The CheckMate 016 Study. J Clin Oncol. 2017 Dec 1;35(34):3851-3858. doi: 10.1200/JCO.2016.72.1985. Epub 2017 Jul 5. PMID 28678668